CLINICAL TRIAL: NCT06033456
Title: Efficacy of Combination of Stellate Ganglion and T2 and T3 Radiofrequency Ablation on Post Mastectomy Complex Regional Pain Syndrome, Randomized Controlled Study.
Brief Title: Combining Stellate Ganglion and T2 and T3 Radiofrequency Ablation on Post-mastectomy Complex Regional Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mary Sabry, Assistant lecturer of Anesthesia, ICU and Pain Management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP2302-301-0001
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Stellate Ganglion; Radiofrequency Ablation; Complex Regional Pain Syndromes; Mastectomy
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Radiofrequency stellate ganglion block using ultrasound guidance (SGB) (Experimental): Visualization of the C6-C7 level will be targeted under fluoroscopic posterior-anterior (PA) guidance. Skin will be infiltrated with 1% lidocaine using a 25-gauge needle. Next, the RF needle will be inserted under a trajectory approach toward the target. Then, with ultrasound guidance, using a superficial linear ultrasound probe to guide further needle penetration so that the needle-tip will lie anterior to the longus colli muscle, the exclusion of vascular structures will be confirmed by duplex.
  Then, 5 to 1 mL of omnipaque dye (iohexol) will be injected. Subsequently, a 100 mm length Baily RF electrode will be inserted and connected to the generator. The RF needle will be positioned alongside the stellate ganglion in the thermal RF technique. With repeated sensory and motor stimulation before RF lesioning .
  Interventions: Procedure: Radiofrequency stellate ganglion block using ultrasound guidance (SGB)
- Radiofrequency thoracic (T2, T3) paravertebral block under fluoroscopic guidance (Experimental): Radiofrequency sympathectomy will be performed with the patient in the prone position. Under fluoroscopic guidance, the T2, T3 vertebral bodies will be identified in an anteroposterior view. For radiofrequency sympathectomy, 10 cm curved, sharp radiofrequency insulated needle with an active tip of 10 mm, needle entry will be performed, and the final placement of the needle tip will be located at the posterior third of the vertebral body in lateral view and just lateral to the body in the anteroposterior view. Once the correct position is confirmed, 0.5 to 1 ml of Omnipaque will be injected, then a 10 cm electrode will be introduced through the RF needle. Before lesioning, a sensory and motor test stimulation is performed to verify the location.
  Interventions: Procedure: Radiofrequency thoracic (T2, T3) paravertebral block under fluoroscopic guidance (TPVB)
- Combined radiofrequency of stellate ganglion block plus thoracic T2, T3 paravertebral block (Experimental): Combination between radiofrequency of stellate ganglion block and thoracic T2, T3 paravertebral block.
  Interventions: Procedure: Combined radiofrequency of stellate ganglion block plus thoracic T2, T3 paravertebral block

INTERVENTIONS:
Procedure: Radiofrequency stellate ganglion block using ultrasound guidance (SGB) — Visualization of C6-C7 level will be targeted under fluoroscopic posterior-anterior (PA) guidance. Skin will be infiltrated with 1% lidocaine using a 25-gauge needle. Next, the RF needle will be inserted under a trajectory approach toward the target. Then, with ultrasound guidance, using a superficial linear ultrasound probe to guide further needle penetration so that the needle-tip will lie anterior to the longus colli muscle, the exclusion of vascular structures will be confirmed by duplex(8).
  Then, 5 to 1 mL of omnipaque dye (iohexol) will be injected. Subsequently, a 100 mm length Baily RF electrode will be inserted and connected to the generator. The RF needle will be positioned alongside the stellate ganglion in the thermal RF technique. With repeated sensory and motor stimulation before RF lesioning
  Arms: Radiofrequency stellate ganglion block using ultrasound guidance (SGB)
Procedure: Radiofrequency thoracic (T2, T3) paravertebral block under fluoroscopic guidance (TPVB) — Radiofrequency sympathectomy will be performed with the patient in the prone position. Under fluoroscopic guidance, the T2, T3 vertebral bodies will be identified in an anteroposterior view. For radiofrequency sympathectomy, 10 cm curved, sharp radiofrequency insulated needle with an active tip of 10 mm, needle entry will be performed, and the final placement of the needle tip will be located at the posterior third of the vertebral body in lateral view and just lateral to the body in the anteroposterior view. Once the correct position is confirmed, 0.5 to 1 ml of Omnipaque will be injected, then a 10 cm electrode will be introduced through the RF needle. Before lesioning, a sensory and motor test stimulation is performed to verify the location.
  Arms: Radiofrequency thoracic (T2, T3) paravertebral block under fluoroscopic guidance
Procedure: Combined radiofrequency of stellate ganglion block plus thoracic T2, T3 paravertebral block — Combination between radiofrequency of stellate ganglion block and thoracic T2, T3 paravertebral block.
  Arms: Combined radiofrequency of stellate ganglion block plus thoracic T2, T3 paravertebral block

SUMMARY:
The aim of this study is to evaluate the efficacy of the combination of Ultra Sound (US) guided radiofrequency stellate ganglion block (SGB) and radiofrequency Thoracic Paravertebral block (TPVB) comparing to US-guided SGB or TPVB alone on the post-mastectomy pain syndrome (PMPS).

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy among females, with an incidence of about 2.1 million women each year. It is the most common cause of cancer-related deaths among women. Modified Radical Mastectomy (MRM) is one of the main surgical treatments for breast cancer. It accounts for 31% of all breast surgery cases. Nearly 40-60% of breast surgery patients experience severe acute postoperative pain, with severe pain persisting for 6-12 months in almost 20-50% of patients (post-mastectomy pain syndrome.

Complex regional pain syndrome (CRPS) is a clinical diagnosis with a highly variable presentation and prognosis. CRPS type I, previously known as reflex sympathetic dystrophy (RSD), is not associated with direct nerve injury. CRPS type II, or causalgia, is associated with direct injury of a specific nerve, often from surgical intervention or trauma. Symptoms include severe pain, sensitivity to light touch, burning, sweating, skin discoloration, edema, temperature changes, loss of motor function, and decreased range of motion of the affected limb. The mechanism of CRPS is not fully understood with central and peripheral sensitization involved.

ELIGIBILITY:
Inclusion Criteria:

* Female patients.
* Type of surgery: Modified Radical Mastectomy MRM.
* Physical status ASA II, III.
* Duration of more than 6 months and less than 2 years.
* Moderate and severe pain (visual analog scale [VAS] ≥ 40 mm).
* Pain described as a refractory to strong opioids (oxycodone) and adjuvant therapy such as(pregabalin) for which more invasive interventions could be tried.

Exclusion Criteria:

* Patient refusal.
* Patient with local and systemic sepsis.
* Local anatomical distortion.
* History of contralateral chest disease or pneumonectomy.
* Known sensitivity or contraindication to the drug used in the study.
* History of psychological disorders.
* Contraindication to regional anesthesia, e.g., pre-existing peripheral neuropathies and coagulopathy.
* Severe respiratory or cardiac disorders. Advanced liver or kidney disease.
* Pregnancy.
* Physical status ASA IV and Male patients.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — * Female patients.
  * Type of surgery: Modified Radical Mastectomy MRM.
Enrollment: 150 (Estimated)
Dates: Start 2023-10-07 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
The degree of pain relief | 3 months after intervention
  Pain relief is assessed by the change in Visual Analogue Scale (VAS) score at 1st day then 1 and 3 months after intervention.
  Complete response VAS 0-3. • Partial response VAS 4-6. • No response VAS 7-10.

SECONDARY OUTCOMES:
Patient satisfaction | 3 months after intervention
  Patient satisfaction by patient satisfaction score (0 very satisfied and 10 dissatisfied)
Oxycodone consumption | 3 months after intervention
  The analgesic concomitant medications (oxycodone) consumption will be assessed prior to the block and at 1st day, 1,3 months.
Pregabalin consumption | 3 months after intervention
  The analgesic concomitant medications (pregabalin) consumption will be assessed prior to the block and at 1st day, 1,3 months.
neuropathic pain | 3 months
  Neuropathic pain will be evaluated according to the Grading System for Neuropathic Pain (GSNP).
  Positive neuropathic cases are those with GSNP 3 (probable) or GSNP 4 (definite) .
  The grading system for neuropathic pain (GSNP) is as follows: Grade 1 (unlikely), Grade 2 (possible), Grade 3 (probable), and Grade 4 (definite)
Patient's Quality of life | 3 months
  Patient's Quality of life according to WHOQOL(who measure quality of life)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: after the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.